CLINICAL TRIAL: NCT05690035
Title: PD-1 Antibody (Tislelizumab) Combined With VEGFR 1/2/3 Inhibitor (Fruquintinib) for ARID1A-mutated Metastatic pMMR/MSS Colorectal Cancer: an Open-label, Multi-center, Phase II Clinical Trial
Brief Title: Tislelizumab Combined With Fruquintinib for Metastatic pMMR/MSS Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow patient recruiting. No patients were enrolled 12 months after study initiation.
Sponsor: Sun Yat-sen University (Other)
Collaborators: Hutchmed (Industry); BeiGene (Industry)
Responsible Party: Principal Investigator, Pei-Rong Ding, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2022-653-01
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Colorectal Cancer; mCRC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tislelizumab; HMPL-013

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with mCRC (Experimental): Tislelizumab 200mg ivdrip every 3 weeks; Fruquintinib 5mg qd day 1-14, every 3 weeks
  Interventions: Drug: Tislelizumab & Fruquintinib

INTERVENTIONS:
Drug: Tislelizumab & Fruquintinib — combinational treatment of Tislelizumab and Fruquintinib until PD, intolerable toxicity, death or withdrawal of informed consent

SUMMARY:
This is an open-label phase II study, with the aim of investigating the efficacy and safety of Tislelizumab + Fruquintinib combination therapy in ARID1A-mutated pMMR/MSS metastatic colorectal cancer who have been treated with standard chemotherapy that includes fluoropyrimidine, oxaliplatin, and irinotecan. Patients with hypermutated CRC that carries POLE/POLD1 mutations cannot be included.

DETAILED DESCRIPTION:
In this open-label phase II study, patients with ARID1A-mutated pMMR/MSS metastatic colorectal cancer who have been treated with standard chemotherapy that includes fluoropyrimidine, oxaliplatin, and irinotecan, will be scheduled for Tislelizumab (200mg ivdrip Q3W day1) + Fruquintinib (5mg/day Q3W day1-14) until intolerable toxicity, disease progression or death. Primary endpoint of this study is ORR and secondary endpoints are OS, PFS, DCR and safety.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old (including 18 and 80);
* Histologically confirmed colorectal adenocarcinoma and biopsy pathology confirmed MSS/pMMR;
* Gene testing confirmed ARID1A gene mutation (nonsynonymous);
* No signs of intestinal obstruction; Or intestinal obstruction has been relieved after proximal colostomy;
* Has received and failed ≥ 2 line of chemotherapy or progressed on or intolerable to oxaliplatin, irinotecan and fluorouracil chemotherapy after diagnosed with mCRC;
* ECOG PS 0-2;
* Able to swallow tablets;
* Life expectancy of greater than 3 months;
* Adequate bone marrow and organ function;
* If female and of childbearing potential, must:
* Have a negative pregnancy test ≤14 days prior to initiating study treatment
* Agree to avoid pregnancy during and for 3 months after study treatment

If male with a partner of childbearing potential, must:

* Agree to use adequate, medically approved, contraceptive precautions during and for 3 months after the last dose of study treatment.
* Able and willing to provide written informed consent for the study.

Exclusion Criteria:

* Any active autoimmune disease or history of autoimmune disease;
* Those who are using immunosuppressive agents, or systemic or absorbable local hormone therapy to achieve immunosuppressive purpose, and continue to use within 2 weeks before enrollment;
* Severe allergic reaction to other monoclonal antibodies;
* Subjects with clinical symptoms of untreated active brain metastasis or meningeal metastasis;
* Have received other PD-1 antibody therapy or other immunotherapy targeting PD-1/PD-L1 in the past;
* Patients with high TMB (≥ 30Muts/Mb) and germline or somatic POLE/POLD1 gene mutations in the exonuclease domain;
* There are clinical symptoms or diseases of heart that are not well controlled, such as: (a) heart failure of NYHA level 2 or above (b) unstable angina pectoris (c) myocardial infarction occurred within 1 year (d) clinically significant supraventricular or ventricular arrhythmia needs treatment or intervention;
* Known hereditary or acquired bleeding and thrombophilia or being treated with thrombolysis or anticoagulation;
* Urinary protein ≥ ++, or the 24-hour urine protein quantification greater than 1.0g;
* Clinically significant bleeding symptoms or clear bleeding tendency within 3 months before enrollment;
* Subjects with active infection;
* Congenital or acquired immune deficiency (such as HIV infected persons), or active hepatitis (hepatitis B: HBsAg positive and HBV DNA ≥ 10^4 copies/ml; hepatitis C: HCV antibody positive);
* Other advanced malignant tumors within 5 years (except cured skin basal cell carcinoma, cervical carcinoma in situ, ovarian cancer, thyroid cancer and breast cancer);
* Live vaccine may be inoculated less than 4 weeks before the study medication or during the study period;
* Known or suspected to be allergic to the study drug or to any drug given in this trial;
* Have any other disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other conditions that makes the subject not eligible according to the judgment of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 3 years
  The proportion of patients with a confirmed complete response or partial response

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | up to 3 years
  PFS is defined as the time from enrollment to the first documented progressive disease (PD) or death due to any cause, whichever occurred first.
Overall Survival (OS) | up to 3 years
  OS is defined as the time from enrollment to death due to any cause.
Disease control rate | up to 3 years
  The proportion of patients with a best overall response of confirmed complete or partial response, or stable disease (CR+ PR + SD).
Incidence of Treatment-Emergent Adverse Events | until 60 days after last patient last study drug treatment
  Safety and tolerance evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Peirong Ding, M.D., Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Sun Yat-sen University, Cancer Center, Guangzhou, Guangdong
  - Xiaoshi Zhang, Guangzhou

IPD SHARING:
Plan to Share IPD: No